CLINICAL TRIAL: NCT02220764
Title: Prospective Evaluation of Zirconia Based Tooth- and Implant- Supported Fixed Dental Prostheses
Brief Title: Zirconia Based Fixed Dental Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W-008
Record Dates: First submitted 2014-07-16; First posted 2014-08-20 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Zirconia Based Fixed Dental Prostheses
Keywords: prospective study; chipping; survival rate; fracture resistance; zirconia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tooth-supported (Experimental): Long-span tooth-supported zirconia based fixed dental prostheses
  Interventions: Device: Teeth abutment
- Implant-supported (Active Comparator): Long-span implant-supported zirconia based fixed dental prostheses
  Interventions: Device: Implant abutments

INTERVENTIONS:
Device: Teeth abutment
  Other Names: Zenotec system
  Arms: Tooth-supported
Device: Implant abutments
  Other Names: Zenotec system; Wital (Implant system)
  Arms: Implant-supported

SUMMARY:
The objective of this prospective clinical study is to investigate the differences in the complication rates between tooth- and implant- supported zirconia based fixed dental prostheses (FDPs) with at least 4 units. The null-hypothesis is that there is no difference in the complication rates between implant- supported and tooth- supported zirconia FDPs.

DETAILED DESCRIPTION:
The study aims to provide evidence regarding the clinical behaviour of long-span tooth- and implant-supported FDPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Missing of at least two adjacent teeth in the maxilla or mandibular
* Sufficient oral hygiene

Exclusion Criteria:

* Addiction to alcohol or drugs
* Severe craniomandibular disorders
* Severe systematic diseases
* Patients unable or unwilling to sign the informed consent form
* Untreated periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

REFERENCES:
- [Derived] Konstantinidis IK, Jacoby S, Radel M, Boning K. Prospective evaluation of zirconia based tooth- and implant-supported fixed dental prostheses: 3-year results. J Dent. 2015 Jan;43(1):87-93. doi: 10.1016/j.jdent.2014.10.011. Epub 2014 Nov 5. PMID 25446240

RESULTS

PARTICIPANT FLOW:
Groups:
- Tooth-supported: Long-span tooth-supported zirconia based fixed dental prostheses
  Teeth abutment
- Implant-supported: Long-span implant-supported zirconia based fixed dental prostheses
  Implant abutments
Period: Overall Study
Arm/Group | Tooth-supported | Implant-supported
Started | 24 | 8
Completed | 20 | 7
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tooth-supported | Implant-supported | Total
Number analyzed (Participants) | 24 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.01) | 53.9 (10.9) | 54.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Fixed Dental Prostheses (FDPs) With Failure
Description: "Failure" was recorded if there was a need to remove the Fixed Dental Prosthesis over the observation period.
Time Frame: 3 years
Measure: Number; unit: FDPs with failure
Arm/Group | Tooth-supported | Implant-supported
Number analyzed (Participants) | 20 | 7
FDPs with failure | 0 | 1

2. Secondary Outcome: Number of Fixed Dental Prostheses (FDPs) With Chip/s
Description: Measurement of the amount of fractures of the veneering material 6,12,18,24,30 and 36 months after placement of the restorations. The percentage of chips for the implant- and tooth- supported restorations will be reported.
Time Frame: 3 years
Measure: Number; unit: FDPs with chip/s
Arm/Group | Tooth-supported | Implant-supported
Number analyzed (Participants) | 20 | 7
FDPs with chip/s | 3 | 5
Statistical Analysis 1: Comparison: Tooth-supported vs Implant-supported; Null hypothesis: The chipping rates between tooth- and implant- supoorted FDPs are equally distributed; Test type: Superiority or Other; p = 0.03, Log Rank

3. Other Pre Specified Outcome: Number of of Fixed Dental Prostheses (FDPs) With Rough Surface
Description: Measurement of the restorations with rough surface 6,12,18,24,30 and 36 months after placement of the restorations.
Time Frame: 3 years
Measure: Number; unit: FDPs with rough surface
Arm/Group | Tooth-supported | Implant-supported
Number analyzed (Participants) | 20 | 7
FDPs with rough surface | 13 | 7

ADVERSE EVENTS:
Arm/Group | Tooth-supported | Implant-supported
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/8
Other Adverse Events (participants affected / at risk) | 0/24 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No